## **Statistical Analysis Plan**

**Study ID: 213352** 

Official Title of Study: Phase 2, Multi-Arm Study of Niraparib Administered Alone and in Combination with a PD1 inhibitor in Patients with Non-Small Cell Lung Cancer

Other Identifiers: 3000-02-001

**Date of Document: 27-AUG-2019** 

# STATISTICAL ANALYSIS PLAN: Study 3000-02-001

**Protocol Title:** Phase 2, Multi-Arm Study of Niraparib Administered

Alone and in Combination with a PD1 inhibitor in Patients

with Non-Small Cell Lung Cancer

**Protocol Number:** 3000-02-001

**Protocol Version and Date:** Version 3.0, 31 May 31 2018 (amendment 2)

Version 2.0, 05 September 2017 (Amendment 1)

Version 1.0, 17 May 2017 (Original)

**Study Phase:** Phase 2

**Product Name:** Niraparib, Pembrolizumab, and TSR-042

**Sponsor:** TESARO, Inc.

**Analysis Plan Version and Date:** Version 0.8, 27 August 2019

#### **Confidentiality Statement**

All information contained in this document is privileged and confidential to TESARO. Any distribution, copying, or disclosure is strictly prohibited without prior written approval by TESARO.

## **SPONSOR SIGNATURES**

**Protocol Title:** Phase 2, Multi-Arm Study of Niraparib Administered Alone and in

Combination with a PD1 inhibitor in Patients with Non-Small Cell Lung

Cancer

**Protocol Number:** 3000-02-001

By signing this document, I acknowledge that I have read the document and approve of the planned statistical analyses described herein. I agree that the planned statistical analyses are appropriate for this study, are in accordance with the study objectives, and are consistent with the statistical methodology described in the protocol, clinical development plan, and all applicable regulatory guidance and guidelines.

#### Author

PPD , PhD Signature:
PPD Date:

LLX Solutions, LLC

#### **Approver:**

Yongqiang Tang, PhD Signature:

Director of Biostatistics Date:

TESARO, Inc.

Iryna Teslenko, MD Signature:

Senior Medical Director, Date:

Clinical Research, TESARO, Inc.

Confidential Page 2 of 45

# **TABLE OF CONTENTS**

| SI | PONSO | R SIGNATURES | 2 |
|---|---|---|---|
| $\mathbf{T}_{A}$ | ABLE ( | OF CONTENTS | 3 |
| Ll | IST OF | ABBREVIATIONS | 6 |
| 1 | INTI | RODUCTION | 8 |
| 2 | STU | DY DESIGN OVERVIEW | 8 |
| | 2.1 | Overall Study Design | 8 |
| | 2.2 | Sample Size | 18 |
| | 2.3 | Randomization and Blinding | 19 |
| 3 | STU | DY OBJECTIVES | 19 |
| | 3.1 | Primary Objectives | 19 |
| | 3.2 | Secondary Objectives | 19 |
| 4 | STU | DY ENDPOINTS AND EVALUATIONS | 20 |
| | 4.1 | Efficacy Endpoints | 20 |
| | 4.1 | .1 Primary Efficacy Endpoint | 20 |
| | 4.1 | .2 Secondary Efficacy Endpoints | 20 |
| | 4.2 | Safety Evaluations | 23 |
| | 4.3 | Other Evaluations | 23 |
| 5 | <b>PLA</b> | NNED ANALYSES | 24 |
| | 5.1 | Changes from planned Analyses in the Protocol | 24 |
| | 5.2 | Interim Analyses | 24 |
| | 5.3 | Final Analyses and Reporting | 24 |
| 6 | ANA | LYSIS POPULATIONS AND APPLICATIONS | 24 |
| | 6.1 | Modified Intent-to-Treat Population | 24 |
| | 6.2 | Pharmacokinetic Population | 24 |
| | 6.3 | Safety Population | 24 |
| | 6.4 | Application of Analysis Populations | 25 |
| 7 | STA | TISTICAL CONSIDERATIONS | 26 |
| | <b>7.1</b> | General Statistical Procedures | 26 |
| | 7.2 | Patient Enrolment and Disposition | 27 |
| | 7.2 | Patient Enrollment | 27 |
| | 7.2 | Patient Disposition | 27 |
| | 7.2 | Protocol Deviations | 27 |
| | 7.3 | Demographic and Other Pre-treatment Variables | 28 |
| | 7.3 | | |
| | _ | History | |
| | 7.3 | J | |
| | 7 3 | 3.3 Medication Use/Procedures | 30 |

| | <b>7.4</b> A | Analysis of Efficacy Data | 31 |
|----|--------------|------------------------------------------------|----|
| | 7.4.1 | Primary Efficacy Data | 31 |
| | 7.4.2 | 2 Secondary Efficacy Data | 32 |
| | <b>7.5</b> A | Analysis of Safety Data | 32 |
| | 7.5.1 | Adverse Events | 32 |
| | 7.5.2 | 2 Study Drug Exposure and Compliance | 34 |
| | 7.5.3 | Clinical Laboratory Evaluations | 36 |
| | 7.5.4 | 4 Vital Signs | 37 |
| | 7.5.5 | 5 Electrocardiogram | 37 |
| | 7.5.6 | 6 Physical Examinations | 38 |
| | 7.5.7 | 7 ECOG Performance Status | 38 |
| 8 | DEFIN | NITIONS AND CONVENTIONS FOR DATA HANDLING | 38 |
| | 8.1 I | Definition of Baseline | 39 |
| | <b>8.2</b> A | Analysis Visit Window | 39 |
| | 8.3 I | Efficacy Data Handling | 39 |
| | 8.4 | Safety Data Handling | 39 |
| | 8.4.1 | Handling of Repeated Clinical Laboratory Tests | 39 |
| | 8.4.2 | 2 Handling of Partial Dates for AEs | 39 |
| | 8.4.3 | Handling of Partial Dates for Medications | 40 |
| 9 | REFE | RENCE | 41 |
| 10 | APPE | NDICES | 42 |

## **TABLES**

| Table 1: Schedule of Events for Cohort 1, 1A, 2, 2A | 11 |
|---|---|
| Table 2: Schedule of Events for Cohort 3 | 15 |
| Table 3: Sample Size by Cohort | 18 |
| Table 4: Criteria for Considering Treatment Efficacious by Cohort and Stage | 19 |
| Table 5: Censoring Rules for DOR | 21 |
| Table 6: Censoring Rules for PFS | 22 |
| Table 7: Application of Analysis Populations for Tables and Graphs | 26 |
| Table 8: RECIST Response for Patients with Measurable Disease | 43 |
| Table 9: Common Terminology Criteria for Adverse Events v4.03 (CTCAE) | 44 |

# **LIST OF ABBREVIATIONS**

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| AE | adverse event |
| AESI | adverse event of special interest |
| ALK | anaplastic lymphoma kinase |
| aPTT | activated partial thromboplastin time |
| AST | aspartate aminotransferase |
| BMI | body mass index |
| BOR | best overall response |
| CI | confidence interval |
| CBC | complete blood count |
| CR | complete response |
| CT | computed tomography |
| CTCAE | common terminology criteria for adverse events |
| ECOG | Easter Cooperative Oncology Group |
| eCRF | electronic case report form |
| EGFR | epidermal growth factor receptor |
| EOS | end of study |
| ЕОТ | end of treatment |
| FDA | US Food and Drug Administration |
| LLN | lower limit of normal |
| MedDRA | medical dictionary for regulatory activities |
| NSCLC | non-small cell lung cancer |
| ORR | objective response rate |
| OS | overall survival |
| PD | progressive disease |
| PD-1 | programmed cell death-1 |
| PD-L1 | programmed death-ligand 1 |
| PFS | progression-free survival |
| PK | pharmacokinetics |
| PO | oral(ly) |

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| PR | partial response |
| PT | preferred term |
| Q1 | first quartile |
| Q3 | third quartile |
| QD | once daily |
| RECIST | response evaluation criteria in solid tumors |
| RRs | standard of care response rate |
| RRt | target response rate |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SOC | system organ class |
| SD | stable disease or standard deviation |
| sqNSCLC | squamous non-small cell lung cancer |
| TEAE | treatment-emergent adverse event |
| TPS | tumor proportion score |
| TSH | thyroid-stimulating hormone |
| ULN | upper limit of normal |
| WHO | World Health Organization |

### 1 INTRODUCTION

This statistical analysis plan (SAP) provide the detailed statistical methods to be used for analyses and data presentation for reporting efficacy, safety, non-compartmental Pharmacokinetics of investigational drug niraparib for TESARO study protocol 3000-02-01.

The pharmacokinetics and exposure-response analyses will be provided in a separate document. The exploration of blood and tumor-based biomarkers that predict sensitivity or resistance to niraparib will also be detailed in a separate document. This document has been prepared according to Study Protocol Amendment 2 dated 31 May 2018.

### 2 STUDY DESIGN OVERVIEW

## 2.1 Overall Study Design

This is a multicenter, open-label, multi-arm Phase 2 study to evaluate the efficacy and safety of single agent niraparib in patients with locally advanced and metastatic squamous non-small cell lung cancer (sqNSCLC) and of the combination of niraparib and a PD-1 inhibitor in locally advanced and metastatic non-small cell lung cancer (NSCLC) all histologies patients.

The study has 2 stages, each of which will evaluate separate cohorts of different cancer patients with a sample size that is deemed statistically significant to determine whether further examination may be warranted in the individual indications. In Stage 1, Cohorts 1 and 2 will receive niraparib plus the PD-1 inhibitor pembrolizumab, and Cohort 3 will receive niraparib alone. In Stage 2, Cohorts 1A and 2A will receive niraparib plus the PD-1 inhibitor TSR-042. The study design is presented graphically in Figure 1.

Figure 1 Study Design

#### Stage 1:



Stage 2:



<sup>\*</sup>Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease

Abbreviations: NSCLC = non-small cell lung cancer; PD-1 = programmed cell death-1;

PD-L1 = programmed death ligand-1; TPS = Tumor Proportion Score

**Cohorts 1 and 1A:** Locally advanced and metastatic NSCLC patients (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment, whose tumors have high PD-L1 expression (TPS ≥ 50%), and no known epidermal growth factor receptor (EGFR) sensitizing mutation and/or ROS-1 or anaplastic lymphoma kinase (ALK) translocations will receive combination of niraparib and a PD-1 inhibitor (pembrolizumab or TSR-042). *Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease.* 

Cohorts 2 and 2A: Locally advanced and metastatic NSCLC patients (all histologies) with no prior systemic chemotherapy or PD-1/PD-L1 inhibitor treatment, whose tumors have PD-L1 expression (TPS between 1% and 49%) and no known EGFR sensitizing mutation and/or ROS-1 or ALK translocations, will receive combination of niraparib and a PD-1 inhibitor (pembrolizumab or TSR-042). Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease.

**Cohort 3:** Locally advanced and metastatic sqNSCLC patients who have been previously treated with both platinum and either PD-1 or PD-L1 inhibitor will receive single agent niraparib.

This study will consist of a Screening Period (Day -21 to Day -1), a Treatment Period, an End of Treatment (EOT) Period occurring within 7 days of the decision to discontinue treatment for any reason, a Safety Follow-up Visit occurring 30 + 7 days after the last dose of study drug, and a Follow-up Assessment occurring every  $90 \pm 14$  days, which will continue until death or the end of study data collection (a minimum of 6 months after the enrollment of the last patient, provided that this allows the opportunity for completion of all 90-day follow-up assessments).

The schedules of assessments for cohorts are presented in Table 1 and Table 2.

Table 1: Schedule of Events for Cohort 1, 1A, 2, 2A

| Screening | | Cycle 1 | | Subsequent<br>Cycles | ЕОТ | Safety<br>Follow-Up | Follow-Up<br>Assessment |
|---|---|---|---|---|---|---|---|
| -21 to -1 | 1 | 8 | 15 | Cycle n,<br>Day 1 | | 30 + 7 days<br>post-treatment | (every 90 ±<br>14 days) |
| X | | | | | | | |
| X | X | | | | | | |
| X | | | | | | | |
| X | | | | | | | |
| $X^1$ | | | | | | | |
| X | | | | $X^2$ | X | | |
| | X | | | | | | |
| | X <sup>3, 4</sup> | | | X <sup>3, 4</sup> | | | |
| X <sup>5</sup> | performedose. Subperformed Week 72 | formed 9 weeks $(63 \pm 7 \text{ days})$ after first<br>e. Subsequent tumor imaging will be<br>formed every 9 weeks $(63 \pm 7 \text{ days})$ until<br>ek 72 and every 12 weeks $(84 \pm 7 \text{ days})$ weeks $(84 \pm 7 \text{ days})$ week 72 and every 12 weeks $(84 \pm 7 \text{ days})$ | | | | th, withdrawal of p, imaging should $3 \pm 7$ days) until | |
| X | X <sup>7</sup> | X | X | X | X | X | X <sup>8</sup> |
| | -21 to -1 X X X X X X | -21 to -1 X X X X X X X X X X X X X | -21 to -1 1 8 X X X X X X X X X X X X | -21 to -1 1 8 15 X X X X X X X X X X X X X | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Cycles -21 to -1 | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ |

| Cycle/Visit | Screening | | Cycle 1 | | Subsequent<br>Cycles | ЕОТ | Safety<br>Follow-Up | Follow-Up<br>Assessment |
|---|---|---|---|---|---|---|---|---|
| Day of Procedure | -21 to -1 | 1 | 8 | 15 | Cycle n,<br>Day 1 | | 30 + 7 days<br>post-treatment | (every 90 ±<br>14 days) |
| Serum chemistry | X | $X^7$ | | X | X | X | X | $X^8$ |
| Pregnancy test <sup>9</sup> | X | | | | | | | |
| Urinalysis | X | | | | | | | |
| TSH, T3 or FT3, and FT4 | $X^{10}$ | | | | X <sup>10</sup> | X <sup>10</sup> | $X^{10}$ | |
| ECG | X | | | | | X | | |
| Physical examination | X | | | | | X | | |
| Symptom-directed physical examination | | X | | X | X | | X | |
| Vital signs and weight | X | X | | | X | X | X | |
| Height | X | | | | | | | |
| ECOG performance status | X | X | | | X | X | | |
| Concomitant medications/procedures <sup>11</sup> | | Re | corded from | first dose o | f study drug throu | gh Safety | Follow-up | |
| AE monitoring <sup>12</sup> | X | X | X | X | X | X | X <sup>13</sup> | X <sup>13</sup> |
| Pembrolizumab treatment administered <sup>14</sup> (Stage 1 only) | | X | | | X | | | |
| TSR-042 treatment administered (Stage 2 only) | | X | | | X <sup>15</sup> | | | |
| Niraparib treatment dispensed/collected | | X | | | X | X | | |
| Survival/AESI (regardless of causality) and study-drug related SAEs | | | | | | | | |

| Cycle/Visit | Screening | Cycle 1 | | Subsequent<br>Cycles | EOT | Safety<br>Follow-Up | Follow-Up<br>Assessment | |
|---|---|---|---|---|---|---|---|---|
| Day of Procedure | -21 to -1 | 1 | 8 | 15 | Cycle n,<br>Day 1 | | 30 + 7 days<br>post-treatment | (every 90 ±<br>14 days) |
| (Telephone assessment allowed) | | | | | | | | X <sup>16</sup> |

Abbreviations: AE = adverse event; AESI = Adverse Event of Special Interest, CBC = complete blood count; CTC = circulating tumor cell; ctDNA = circulating tumor DNA; DNA = deoxyribonucleic acid; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; EOT = end of treatment; FFPE = formalin fixed paraffin embedded; FT3 = free triiodothyronine; FT4 = free thyroxine; ICF = informed consent form; PK = pharmacokinetics; RECIST = Response Evaluation Criteria in Solid Tumors; SAE = serious adverse event; T3 = triiodothyronine; TSH = thyroid-stimulating hormone.

- <sup>1</sup> An archival FFPE tumor tissue specimen, which may have been collected at any time prior to Screening, should be submitted for exploratory biomarker analysis within 30 days of the patient's first dose. If no archival FFPE tumor tissue is available, a tumor tissue biopsy should be obtained before Cycle 1/Day 1.
- <sup>2</sup> Required for Cycle 2/Day 1 only.
- <sup>3</sup> Blood sample for niraparib and pembrolizumab PK will be collected on Cycle 1/Day 1, Cycle 2/Day 1, Cycle 4/Day1, and Cycle 8/ Day 1 (or EOT if patient discontinues before Cycle 8) in all patients in Cohorts 1 and 2. Blood samples for PK assessment of niraparib will be collected in Cycle 1/Day 1, Cycle 2/Day 1, Cycle 4/Day 1, and Cycle 9/Day 1 (or EOT if patient discontinues before Cycle 9) in all patients in Cohorts 1A and 2A. Blood sample for TSR-042 will be collected on Cycle 1/Day 1, Cycle 2/Day 1, Cycle 4/Day1, and Cycle 9/ Day 1 (or EOT if patient discontinues before Cycle 9). See Table 15 of protocol for detailed schedule.
- <sup>4</sup> Intensive niraparib PK sampling will be collected only for a subset of patients (N = 8/cohort) in Cycle 1 and Cycle 4. See Section 8.3 and Table 16 of protocol for detailed schedule. Patients in this subset will be instructed to hold their niraparib dose, which will be taken in clinic on specified days for PK sampling.
- <sup>5</sup> Scans performed prior to the signing of the ICF as part of routine clinical management are acceptable for use as initial tumor imaging if they are of diagnostic quality and are performed within 28 days prior to first dose date
- <sup>6</sup> For details on tumor assessment per RECIST v1.1 see Section 7.3.1, Section 8.2, and Appendix C of protocol. All radiographic images/scans at the specified time points as well as any unscheduled images/scans should be archived by the study sites for potential future evaluation.
- <sup>7</sup> If screening assessments were performed within 72 hours of Day 1, repeat testing is not required.
- <sup>8</sup> CBC and serum chemistry at the Follow-up Assessment should be conducted only on Day 90 post-treatment to assess for possible AESI (Section 7.1.6 of protocol).
- <sup>9</sup> Serum pregnancy test for women of childbearing potential within 72 hours of first dose of study treatment. If the serum pregnancy result is not available before dosing, a urine pregnancy test may be performed.
- <sup>10</sup>Blood samples for TSH, T3 or FT3, and FT4 are to be collected at screening, every 6 weeks from Cycle 1/Day 1, and at EOT. Blood samples for TSH, T3 or FT3, and FT4 should be collected at 30-day post-treatment Safety Follow-up only if assessment is clinically indicated.
- <sup>11</sup>Any new anticancer treatment started during the study should also be collected.

| Cycle/Visit | Screening | Cycle 1 | | | Subsequent<br>Cycles | ЕОТ | Safety<br>Follow-Up | Follow-Up<br>Assessment |
|---|---|---|---|---|---|---|---|---|
| Day of Procedure | -21 to -1 | 1 | 8 | 15 | Cycle n,<br>Day 1 | | 30 + 7 days<br>post-treatment | (every 90 ±<br>14 days) |

<sup>&</sup>lt;sup>12</sup>Collection of AEs begins when the ICF is signed.

<sup>&</sup>lt;sup>13</sup>AEs are required to be captured through 30 days after cessation of study treatment (Section 7.1.3 of protocol). However, SAEs are required to be captured through 90 days after cessation of study treatment (or to a minimum of 30 days post-treatment if the patient starts alternate anticancer therapy) (Section 7.1.5 of protocol), and any pregnancies that occur within 180 days post-treatment are to be captured. AESIs should be collected until study closeout, regardless of causality (Section 7.1.6 of protocol).

<sup>&</sup>lt;sup>14</sup>Pembrolizumab should be administered once every 21 days (200 mg intravenous) on Day 1 of each cycle. Pembrolizumab may be administered up to 3 days before or after the scheduled Day 1 of each cycle after Cycle 1 due to administrative reasons. On days where pembrolizumab is administered, it should be administered before niraparib.

<sup>&</sup>lt;sup>15</sup>TSR-042 will be administered at a dose of 500 mg on Day 1 every 3 weeks in Cycles 1 through 4, followed by 1,000 mg every other cycle (every 6 weeks) thereafter, beginning on Cycle 5 Day 1. On days where TSR-042 is administered, it should be administered before niraparib.

<sup>&</sup>lt;sup>16</sup>Patients will be followed until study closeout for survival status, AESI (regardless of causality), and study-drug related SAEs (Section 7.1.6 of protocol).

Table 2: Schedule of Events for Cohort 3

| Cycle/Visit: | Screening | | Cycle 1 | | Subsequent<br>Cycles | ЕОТ | Safety<br>Follow-Up<br>30 + 7 days<br>post-treatment | Follow-Up<br>Assessment<br>(every 90 ± 14<br>days) |
|---|---|---|---|---|---|---|---|---|
| Day of Procedure | -21 to -1 | 1 | 8 | 15 | Cycle n,<br>Day 1 | | | |
| Informed consent | X | | | | | | | |
| Inclusion/exclusion criteria review | X | X | | | | | | |
| Demographics | X | | | | | | | |
| Medical, surgical, cancer, smoking, and medication history | X | | | | | | | |
| Archival tumor tissue | $X^1$ | | | | | | | |
| Blood sample for ctDNA | X | | | | X <sup>2</sup> | X | | |
| Blood sample for CTC | | X | | | | | | |
| Blood sample for PK | | X <sup>3, 4</sup> | | | X <sup>3, 4</sup> | | | |
| Tumor assessment | X <sup>5</sup> | performe<br>dose. Sub<br>performe<br>Week 24<br>imaging v<br>(63 ± 7 d. | d 6 weeks<br>osequent to<br>d every 6<br>(6 months<br>will be per<br>ays) until | (42 ± 7 day<br>umor imagin<br>weeks (42 ±<br>s). After We<br>formed eve | ± 7 days) until<br>eek 24, tumor<br>ery 9 weeks<br>2 months) and | If patient discontinues treatment for a reason other than progression, death, withdrawal of consent, or loss to follow-up, imaging should continue every 6 weeks (42 ± 7 days) until Week 24 (6 months), then every 9 weeks (63 ± 7 days) until Week 52 (12 months) and every 12 weeks (84 ± 7 days) thereafter <sup>6</sup> | | |
| Clinical laboratory assessments | | | | | | | | |
| CBC | X | X <sup>7</sup> | X | X | X | X | X | $X^8$ |
| Serum chemistry | X | $X^7$ | | X | X | X | X | $X^8$ |
| Pregnancy test <sup>9</sup> | X | | | | | | | |
| Urinalysis | X | | | | | | | |
| ECG | X | | | | | X | | |
| Physical examination | X | | | | | X | | |

| Cycle/Visit: | Screening | | Cycle 1 | | Subsequent<br>Cycles | ЕОТ | Safety<br>Follow-Up | Follow-Up<br>Assessment |
|---|---|---|---|---|---|---|---|---|
| Day of Procedure | -21 to -1 | 1 | 8 | 15 | Cycle n,<br>Day 1 | | 30 + 7 days<br>post-treatment | (every 90 ± 14<br>days) |
| Symptom-directed physical examination | | X | | X | X | | X | |
| Vital signs and weight | X | X | | | X | X | X | |
| Height | X | | | | | | | |
| ECOG performance status | X | X | | | X | X | | |
| Concomitant medications/procedure <sup>10</sup> | | Reco | orded from | first dose | of study drug thro | ugh Safet | ty Follow-up | |
| AE monitoring <sup>11</sup> | X | X | X | X | X | X | X <sup>12</sup> | X <sup>12</sup> |
| Niraparib treatment dispensed/collected | | X | | | X | X | | |
| Survival/AESI (regardless of causality) and study-drug related SAEs (telephone assessment allowed) | | | | | | | | X <sup>13</sup> |

Abbreviations: AE = adverse event; AESI = Adverse Event of Special Interest; CBC = complete blood count; CTC = circulating tumor cell;

DNA = deoxyribonucleic acid; ctDNA = circulating tumor DNA; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; EOT = end of treatment; FFPE = formalin fixed paraffin embedded; ICF = informed consent form; PK = pharmacokinetics; RECIST = Response Evaluation Criteria in Solid Tumors; SAE = serious adverse event

<sup>&</sup>lt;sup>1</sup> An archival FFPE tumor tissue specimen, which may have been collected at any time prior to Screening, should be submitted for exploratory biomarker analysis within 30 days of the patient's first dose. If diagnosis was made by cytology and archival FFPE tissue is not available, patient will not need to provide tumor tissue.

<sup>&</sup>lt;sup>2</sup> Required for Cycle 2/Day 1 only.

<sup>&</sup>lt;sup>3</sup> Blood sample for niraparib PK will be collected on Cycle 1/Day 1, Cycle 2/Day 1, Cycle 4/Day 1, and Cycle 8/Day 1 (or EOT if patient discontinues before Cycle 8). See Table 15 of protocol for detailed schedule.

<sup>&</sup>lt;sup>4</sup> Intensive niraparib PK sampling will be collected only for a subset of patients (N = 8/cohort) on Cycle 1 and Cycle 4. See Section 8.3 and Table 16 of protocol for detailed schedule. Patients in this subset will be instructed to hold their niraparib dose, which will be taken in clinic on specified days for PK sampling.

<sup>&</sup>lt;sup>5</sup> Scans performed prior to the signing of the ICF as part of routine clinical management are acceptable for use as initial tumor imaging if they are of diagnostic quality and are performed within 28 days prior to first dose date.

<sup>&</sup>lt;sup>6</sup> For details on tumor assessment per RECIST v1.1 see Section 7.3.1, Section 8.2 and Appendix C of protocol. All radiographic images/scans at the specified time point as well as any unscheduled images/scans should be archived by the study sites for potential future evaluation.

<sup>&</sup>lt;sup>7</sup> If screening assessments were performed within 72 hours of Day 1, repeat testing is not required.

| Cycle/Visit: | Screening | Cycle 1 | | | Subsequent<br>Cycles | EOT | Safety<br>Follow-Up | Follow-Up<br>Assessment |
|---|---|---|---|---|---|---|---|---|
| Day of Procedure | -21 to -1 | 1 | 8 | 15 | Cycle n,<br>Day 1 | | 30 + 7 days<br>post-treatment | (every 90 ± 14<br>days) |

<sup>&</sup>lt;sup>8</sup> CBC and serum chemistry at the Follow-up Assessment should be conducted only on Day 90 post-treatment to assess for possible AESI (Section 7.1.6 of protocol)

<sup>&</sup>lt;sup>9</sup> Serum pregnancy test for women of childbearing potential within 72 hours of first dose of study treatment. If the serum pregnancy result is not available before dosing, a urine pregnancy test may be performed.

<sup>&</sup>lt;sup>10</sup> Any new anticancer treatment started during the study should also be collected.

<sup>&</sup>lt;sup>11</sup> Collection of AEs begins when the ICF is signed.

<sup>&</sup>lt;sup>12</sup> AEs are required to be captured through 30 days after cessation of study treatment (Section 7.1.3 of protocol). However, SAEs are required to be captured through 90 days after cessation of study treatment (or to a minimum of 30 days post-treatment if the patient starts alternate anticancer therapy) (Section 7.1.5 of protocol), and any pregnancies that occur within 180 days post-treatment are to be captured. AESIs should be collected until study closeout, regardless of causality (Section 7.1.6 of protocol).

<sup>&</sup>lt;sup>13</sup> Patients will be followed until study closeout for survival status, AESI (regardless of causality), and study-drug related SAEs (Section 7.1.6 of protocol).

## 2.2 Sample Size

The null hypothesis for this study is H0:  $ORR \le Standard$  of Care Response Rate (RRs) vs. the alternative hypothesis:  $ORR \ge Target$  Response Rate (RRt) for all cohorts. RRs and RRt for each cohort are specified in Table 3 below.

As different study drugs will be used in Stage 1 and Stage 2, the sample size for each stage was calculated separately for Cohort 1 and Cohort 2. Sample size calculation was based on the primary efficacy endpoint ORR for each cohort assuming a 1-sided alpha level of 0.10 and 80% power.

For Cohorts 1, 2, and 3, the number of patients in Stage 1 was determined based on Simon's 2-stage design. The sample size for Stage 2 (Cohorts 1A and 2A) was calculated based on a 1-stage design. Once enrollment for Stage 1 is completed, Stage 2 enrollment will start. Stage 1 data will be used to determine if further enrollment for Stage 2 is warranted. (Following a cross-program review and decision to move forward with other studies, the Sponsor has decided that Cohort 3 will close to any further enrollment as of Protocol Amendment 2.) The total sample size for this study will range from 59 to 142.

The criteria for rejecting the alternative hypothesis and declaring the experiment treatment as not efficacious at the end of Stage 1 and Stage 2 are listed in Table 4 below. For each cohort, if the number of responders by the end of Stage 1 is the same or less as defined by the criterion, the cohort will be terminated. For a cohort that proceeds to Stage 2, if the total number of responders by the end of Stage 2 is the same or less than the criterion, the alternative hypothesis will be rejected and the experimental treatment will be considered not efficacious for the indication in the cohort, unless the clinical judgment suggests otherwise.

Table 3: Sample Size by Cohort

| | | | | Sample Size | | |
|---|---|---|---|---|---|---|
| Cohort<br>No. | Cohort Description | Target<br>RR | SoC<br>RR | 1st<br>Stage | 2 <sup>nd</sup><br>Stage | Total |
| 1/1A | NSCLC (chemotherapy-naïve, PD-L1 TPS ≥ 50%) | 65% | 45% | 16 | 36 | 52 |
| 2/2A | NSCLC (chemotherapy-naïve, PD-L1 TPS 1-49%) | 50% | 33.5% | 20 | 47 | 67 |
| 3 | SqNSCLC: Platinum and PD-1/PD-L1- treated | 20% | 9% | 23 | 0 | 23 |

Abbreviations: NSCLC = non-small cell lung cancer; PD-1 = programmed cell death-1; PD-L1 = programmed death ligand-1; RR = response rate; SoC = standard of care; SqNSCLC = squamous non-small cell lung cancer; TPS = tumor proportion score.

Table 4: Criteria for Considering Treatment Efficacious by Cohort and Stage

| Cohort<br>No. | Cohort Description | Stage 1<br>Criteria* | Stage 2 Criteria* |
|---|---|---|---|
| 1/1A | NSCLC (chemotherapy-naïve, PD-L1 TPS ≥ 50%) | 8 | 20‡ |
| 2/2A | NSCLC (chemotherapy-naïve, PD-L1 TPS 1-49%) | 7 | 20‡ |
| 3 | SqNSCLC: Platinum and PD-1 or PD-L1-treated | 2 | NA |

Abbreviations: NA = not applicable; NSCLC = non-small cell lung cancer; PD-1 = programmed cell death-1; PD-L1 = programmed death ligand-1; SqNSCLC = squamous non-small cell lung cancer; TPS = tumor proportion score. \* Number of patients with responses (CR/PR) ‡ Not including stage 1 responders.

## 2.3 Randomization and Blinding

This is an open-label study and patients will not be randomized.

## 3 STUDY OBJECTIVES

## 3.1 Primary Objectives

The primary objectives of this study are:

- To evaluate the efficacy of the combination of niraparib and a PD-1 inhibitor in chemotherapy-naïve and PD-1 inhibitor-naïve patients with locally advanced and metastatic NSCLC whose tumors have high PD-L1 expression (TPS ≥ 50%), as assessed by objective response rate (ORR)
- To evaluate the efficacy of the combination of niraparib and a PD-1 inhibitor in chemotherapy-naïve and PD-1inhibitor-naïve patients with locally advanced and metastatic NSCLC whose tumors express PD-L1 (TPS between 1 and 49%) as assessed by ORR
- To evaluate the efficacy of single agent niraparib in patients with metastatic sqNSCLC who have been previously treated with both platinum-based chemotherapy and either PD-1 or PD-L1 inhibitor, as assessed by ORR

# 3.2 Secondary Objectives

The secondary objectives of the study are as follows:

• To evaluate the safety and tolerability of single agent niraparib and of the combination of niraparib and a PD-1 inhibitor

- To evaluate the following additional measures of clinical benefit of single agent niraparib and of the combination of niraparib and a PD-1 inhibitor:
  - o Disease control rate (DCR)
  - o Duration of response (DOR)
  - o Progression-Free Survival (PFS)
  - Overall Survival (OS)

#### 4 STUDY ENDPOINTS AND EVALUATIONS

## 4.1 Efficacy Endpoints

## 4.1.1 Primary Efficacy Endpoint

The primary efficacy endpoint is objective response rate (ORR), defined as the proportion of patients with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) in the analysis population (See Section 6). Tumor assessments after the initiation of further anticancer therapy are excluded for the assessment of BOR.

Response to treatment will be determined based on investigator evaluation of radiographic images according to RECIST v1.1. If CR or PR is observed, tumor imaging for confirmation of response needs to be performed at the earliest 28 days after the first indication of response, but no later than 35 days after the response.

Confirmed BOR will be determined based on the RECIST v1.1. For a confirmed response, the tumor assessment date for the first recorded CR or PR will be considered as the date CR/PR achieved.

All final efficacy analyses for response rate will be based on the confirmed response. Confirmation of response is not required for the purpose of determining if the study should continue enrolling stage 2 patients.

## 4.1.2 Secondary Efficacy Endpoints

#### 4.1.2.1 Disease Control Rate

Disease control rate (DCR) is defined as the proportion of patients with a best overall response of CR, PR or SD.

#### 4.1.2.2 Duration of Response

Duration of Response (DOR) is defined as the time from first documented CR or PR until the subsequently documented disease progression or death, whichever occurs earlier.

DOR will be calculated as shown below for responders only using the censoring rules specified in Table 5.

$$DOR (months) = \frac{\text{Date of PD/Death/Censoring - Date of First recorded CR or PR} + 1}{30.4375}$$

Table 5: Censoring Rules for DOR

| Situation | Date of Event Censoring | Outcome |
|---|---|---|
| Start of subsequent anti-cancer therapy prior to a documented radiologic progression or death | Date of last radiologic tumor assessment prior to or on the date of initiation of the subsequent anti-cancer therapy | Censored |
| No documented radiologic progression, no subsequent anti-cancer therapy started, and no death | Date of last radiologic tumor assessment | Censored |
| Documented radiologic progression or death after<br>two or more consecutive missing radiologic<br>assessments* | Date of last radiologic tumor assessment before the missed tumor assessments | Censored |
| Documented radiologic progression or death without two or more consecutive missing radiologic assessments* | Earliest date of documented radiologic progression or death | Event |

<sup>\*</sup> Cohort 1, 1A, 2, and 2A: On-study tumor imaging requires an assessment every 9 weeks  $(63 \pm 7 \text{ days})$  until Week 72, every 12 weeks  $(84 \pm 7 \text{ days})$  after Week 72 from start of protocol treatment until progression or start of subsequent anticancer treatment.

#### 4.1.2.3 Progression Free Survival (PFS)

PFS defined as the time from the date of first dose to the date of disease progression or death due to any cause, whichever occurs earlier.

PFS will be calculated as shown below using the censoring rules specified in Table 6.

$$PFS(months) = \frac{\text{Date of PD/Death/Censoring - Date of First Dose} + 1}{30.4375}$$

Cohort 3: On-study tumor imaging requires assessment every 6 weeks  $(42 \pm 7 \text{ days})$  until Week 24; every 9 weeks  $(63 \pm 7 \text{ days})$  after Week 24 until Week 52, and then every 12 weeks  $((84 \pm 7 \text{ days}))$  from start of protocol treatment until progression or start of subsequent anticancer treatment.

Table 6: Censoring Rules for PFS

| Situation | Date of Event Censoring | Outcome |
|---|---|---|
| No baseline tumor assessments | First dose date | Censored |
| No post-baseline tumor assessments and no death | First dose date | Censored |
| Start of subsequent anti-cancer therapy prior to a documented radiologic progression or death | Date of last radiologic tumor assessment prior to or on the date of initiation of the subsequent anti-cancer therapy | Censored |
| No documented radiologic progression, no subsequent anti-cancer therapy started, and no death | Date of last radiologic tumor assessment | Censored |
| Documented radiologic progression or death after<br>two or more consecutive missing radiologic<br>assessments* | Date of last radiologic tumor assessment before the missed tumor assessments | Censored |
| Documented radiologic progression or death without two or more consecutive missing radiologic assessments* | Earliest date of documented radiologic progression or death | Event |

<sup>\*</sup> Cohort 1, 1A, 2, and 2A: On-study tumor imaging requires an assessment every 9 weeks  $(63 \pm 7 \text{ days})$  until Week 72, every 12 weeks  $(84 \pm 7 \text{ days})$  after Week 72 from start of protocol treatment until progression or start of subsequent anticancer treatment.

Cohort 3: On-study tumor imaging requires assessment every 6 weeks  $(42 \pm 7 \text{ days})$  until Week 24; every 9 weeks  $(63 \pm 7 \text{ days})$  after Week 24 until Week 52, and then every 12 weeks  $((84 \pm 7 \text{ days}))$  from start of protocol treatment until progression or start of subsequent anticancer treatment.

#### 4.1.2.4 Overall Survival

Overall survival (OS) is defined as the time from date of first dose to the date of death due to any cause. Patients without documented death at the time of the final analysis will be censored at the last known alive date.

The date of last known alive date will be derived for patients not known to have died at the analysis cut-off date using the latest complete date among the following:

- Patient assessment dates (blood sampling [laboratory], vital signs, ECGs, tumor assessment)
- Start and end date of AEs
- Start and end date of study treatment
- Start and end date of subsequent anti-cancer therapies administered after study treatment discontinuation
- Date of study discontinuation for reasons other than lost-to-follow-up
- Last date of contact recorded on the survival follow-up
- Any assessment date after the analysis cut-off date will not be applicable.

OS will be calculated as:

$$OS(months) = \frac{\text{Date of Death/Censoring - Date of First Dose } + 1}{30.4375}$$

## 4.2 Safety Evaluations

The safety evaluations include:

- Treatment emergent adverse events (TEAEs)
- Extent of exposure
- Clinical laboratory assessments
  - Hematology (including CBC and coagulation)
  - Chemistry (including thyroid function tests)
  - Urinalysis
- Serum or urine pregnancy testing
- Vital signs
- Physical examination findings
- ECG

## 4.3 Other Evaluations

Other evaluations include:

- Demographics and baseline characteristics (including NSCLC History)
- Medical history
  - General medical history
  - Other cancer History
  - Surgical history
  - Prior blood disorders
  - Smoking history
- Medication use/procedures
  - Prior medications and concomitant medications
  - Prior anticancer treatment for primary cancer
  - Subsequent anticancer treatment for primary cancer
  - Growth factors
  - Transfusions
  - Concomitant Procedures
  - Concomitant radiotherapy
- ECOG Performance status
- Drug accountability (Niraparib)
- Pembrolizumab Administration

- TSR-042 Administration
- Niraparib dose modification

## 5 PLANNED ANALYSES

## 5.1 Changes from planned Analyses in the Protocol

## 5.2 Interim Analyses

Confirmation of response is not required for the purpose of determining if the study should continue enrolling stage 2 patients. Therefore, there will be no formally interim conducted for the study

## 5.3 Final Analyses and Reporting

All final planned analyses per protocol and this SAP will be performed after database lock. All final efficacy analyses for response rate will be based on the confirmed response.

## 6 ANALYSIS POPULATIONS AND APPLICATIONS

Statistical analysis and data tabulation will be performed using the following analysis populations unless specified otherwise:

## 6.1 Modified Intent-to-Treat Population

Modified intent-to-treat (mITT) population includes all patients who received any study drug and did not withdraw consent prior to having at least one post-baseline tumor assessment. The modified ITT population will be the primary analysis population for the efficacy analyses.

## 6.2 Pharmacokinetic Population

Pharmacokinetic (PK) population includes patients who have at least one of measurable niraparib concentration.

## 6.3 Safety Population

Safety population includes patients who receive at least one dose of either study medications. The safety population will be the primary analysis population for the safety analyses.

## 6.4 Application of Analysis Populations

The analysis population(s) that will be used for creating the summary table(s) of each type is provided in Table 7. All data will be presented in listings for the Enrolled population. A patient will be considered enrolled when the patient has been consented, screened, and all eligibility criteria have been confirmed in the electronic case report form (eCRF).

| Туре | Safety | mITT | PK* |
|--------------------------------------------|--------|------|-----|
| Disposition | X | | X |
| Demographics and baseline characteristics | X | X | |
| Protocol deviations | X | | |
| Medical and disease history | X | | |
| Prior and concomitant medications | X | | |
| Summary and analyses on efficacy endpoints | | X | |
| Summary statistics on PK | | | |
| Safety evaluations | X | | |
| Extent of Exposure | X | | |

Table 7: Application of Analysis Populations for Tables and Graphs

#### 7 STATISTICAL CONSIDERATIONS

All analyses described in this plan are considered priori analyses in that they have been defined prior to locking the database. All other analyses, if any, designed subsequently to locking the database, will be considered post hoc analyses and will be described as exploratory analyses in the Clinical Study Report.

All summaries and analyses for demographics, baseline characteristics, and safety data will be done by cohort and overall separately for

- Stage 1 Receiving Combination of Niraparib and Pembrolizumab
- Stage 1 Receiving Niraparib only Treatment
- Stage 2 Receiving Combination of Niraparib and TSR-042

The summaries and analyses of efficacy data will be provided by stage and cohort.

All summaries and statistical analyses will be performed by SAS v9.3 or later.

#### 7.1 General Statistical Procedures

The descriptive statistics for continuous variables will be the mean, median, standard

<sup>\*</sup> The PK analyses will be provided in a separate document.

deviation (SD), quartiles (Q1, Q3), minimum, maximum, and number of patients.

Frequency distributions for all categorical variables will be presented using counts and percentages.

## 7.2 Patient Enrolment and Disposition

#### 7.2.1 Patient Enrollment

Number of patients will be provided for each analysis population. The denominators for percentages are number of enrolled. A patient is considered as enrolled when the patient has been consented, screened, and all eligibility criteria have been confirmed in the electronic case report form (eCRF).

Enrollment information will be provided in a data listing.

## 7.2.2 Patient Disposition

Patient disposition will be summarized for the Safety population. The summary will present frequency distribution for patients completing the study and discontinuing from the study overall and by reason for discontinuation.

Additionally, the frequency distribution will be provided by reason for discontinuation as applicable for each cohort

- for patients discontinuing treatment niraparib
- for patients discontinuing treatment pembrolizumb
- for patients discontinuing treatment TSR-042

The denominators for calculating the percentages will be based on number of patients for each cohort and overall in the Safety population.

Patient disposition will be provided in a data listing.

#### 7.2.3 Protocol Deviations

A protocol deviation (PD) is any failure to comply with the study protocol as approved by the relevant regulatory authority, ethics committee and/or institutional review board, whether planned or unplanned.

PD will be assessed and classified as important or significant. A protocol deviation is classified as an important PD if there is the potential to:

• Impact the completeness, accuracy, and/or reliability of the study data, or

• Affect a subject's rights, safety, or well-being.

Important protocol deviations require review to confirm whether they are significant. The following are PDs that will always be considered important according to TESARO SOP 1000-00021-CLN:

- Failure to obtain informed consent for participation in the clinical trial
- Enrollment of ineligible subject
- Subject developed withdrawal criteria during the study but was not withdrawn
- Subject received incorrect treatment
- Incorrect or non-compliant dosing of a subject, i.e. dosing that is inconsistent with the protocol
- Administration of an excluded concomitant treatment to a trial subject
- Incorrect cohort assignment

A protocol deviation is classified as a significant PD if it has been confirmed to:

- Adversely impact the completeness, accuracy, and/or reliability of the study data
- Affect a subject's rights, safety, or well-being.

The TESARO medical monitor in conjunction with other study team members as appropriate may determine any PD not listed above to be important or significant based on his/her assessment of (potential) impact. Additionally, a PD could be "downgraded." In this case, the rationale for the change should be documented by the TESARO medical monitor.

Criteria for important and/or significant PDs may be updated as needed throughout the course of the clinical trial.

All PDs will be identified and finalized prior to database lock.

Number and percentage of patients with important or significant protocol deviations will be summarized, further by type of deviation. The denominators for calculating the percentages will be based on number of patients.

All protocol deviations will be listed.

## 7.3 Demographic and Other Pre-treatment Variables

7.3.1 Demographics/Baseline Characteristics and Non-small Cell Lung Cancer History

#### 7.3.1.1 Demographics/Baseline Characteristics

Patient demographics and baseline characteristics include:

- Age (years) calculated as (date of screening date of birth) / 365.25 if date of birth is reported, or age as reported on the eCRF will be used
- Age categories (18 to <65, 65 to <75,  $\ge$ 75; and  $\ge$ 65)
- Race (American Indian/Alaska Native, Asian, Black or African American, Native Hawaiian or other Pacific Islander, White, and Other)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Not Reported, and Unknown)
- Baseline weight (in kilograms; if weight is reported in pounds, convert to kilograms by dividing by 2.2)
- Baseline height (in centimeters; if height is reported in inches, convert to centimeters by multiplying by 2.54)
- Baseline body mass index (BMI) (kg/m2), calculated using the patient's height and weight [BMI (kg/m2) = weight (kg) / height (m)2]
- ECOG performance status at baseline
- Smoking status (Current Smoker, Former Smoker, Never Smoked, Unknown)
- If female, childbearing status (Childbearing potential, Non-childbearing potential)

Continuous data will be summarized for both Safety and mITT populations, using descriptive statistics.

Categorical data will be summarized with frequency distributions using counts and percentages of patients in each category. The denominators for calculating the percentages will be based on the number of patients in both Safety and mITT populations.

Demographics and baseline characteristics will be provided in a listing.

## 7.3.1.2 Non-small Cell Lung Cancer Disease History

The following NSCLC disease history will be collected.

- date of original diagnosis
- overall cancer stage of original diagnosis
- date of first diagnosis of advanced or recurrent or metastatic disease
- stage of first advanced or recurrent or metastatic disease
- histology at diagnosis
- EGFR mutation, KRAS mutation, BRAF mutation, BRCA1/BRCA2 mutation, ALK translocation, and ROS1 translocation.

Time from original diagnosis and time from first diagnosis of advanced or recurrent or metastatic disease to the date of first dose, stages of cancer, histology, mutations and translocations will be summarized using descriptive statistics for continuous variables and frequency distribution for categorical variables.

A data listing will be provided for NSCLC history.

#### 7.3.1.3 PD-L1 Test Results

The PD-L1 test results will be summarized for location of testing, PD-L1 IHC assay, and PD-L1 status as collected on CRF, and percent of TPS.

The PD-L1 test results will be provided data listings.

#### 7.3.2 Medical History

#### 7.3.2.1 General Medical History

The medical history will be coded using the current version of the Medical Dictionary for Regulatory Activities (MedDRA). The frequency count and percentage of patients experiencing any medical conditions will be tabulated by MedDRA SOC and PT for each analysis population. The denominators for calculating the percentages will be based on number of patients in the Safety population.

A data listing of medical history will be provided.

#### 7.3.2.2 Other Cancer History, Surgery History, and Prior Blood Disorders

Prior blood disorders will be coded using current version of MedDRA and summarized by MedDRA SOC, PT and CTCAE grade. Additionally, they will also be summarized by event collected on CRF and CTCAE grade.

Other cancer history will be summarized by the types listed on the CRF as well.

Data listings will be provided separately for other cancer history, surgery, and prior blood disorders.

#### 7.3.3 Medication Use/Procedures

All medications will be coded using the current version of World Health Organization (WHO) Drug Dictionary (WHO-DD). The count and percentage of patients who took prior/concomitant medications will be provided using therapeutic class and WHO Drug preferred name. The denominators for calculating percentages will be based on the number of patients in each cohort of the Safety population. For the summary tables, if a patient has taken a prior or concomitant medication/subsequent treatment more than once, the patient

will be counted only once for the medication/treatment.

Prior medications are defined as medications received prior to the first dose of either study drugs. Concomitant medications are defined as medications received during the treatment period.

Prior and subsequent anticancer treatments for primary cancer will be summarized for the following information:

- agent name listed on CRF
- reason for administration
- number of anticancer treatments (categorical)
- number of anticancer treatments (categorical) in neoadjuvant, adjuvant, metastatic and other settings
- time since the end of last anticancer treatment (months)
- best response of last anticancer treatment
- reason for discontinuation
- treatment ongoing (only for subsequent)

The denominators for calculating the percentages will be based on number of patients in each cohort of safety population.

Number of patients receiving transfusions will be summarized by the type of transfusions. For each type of transfusion, number of units transfused will be presented in the table.

All medications, prior and subsequent anticancer treatments, and transfusions will be provided in data listings. In addition, separate listings will be provided for:

- Growth factors
- Concomitant Procedures
- Concomitant radiotherapy

## 7.4 Analysis of Efficacy Data

## 7.4.1 Primary Efficacy Data

The primary efficacy variable is objective response rate (ORR), defined as the proportion of patients with a confirmed best overall response of complete response (CR) or partial response

(PR) in the analysis population. Tumor assessments after the initiation of further anticancer therapy are excluded for the assessment of best overall response.

Number of responders, ORR, and its two-sided 80% and 95% binomial exact (Clopper-Pearson) confidence interval will be reported for each cohort.

## 7.4.2 Secondary Efficacy Data

DCR will be analyzed using the same methods for ORR for each cohort.

For each cohort, time-to-event variables (DOR, PFS, and OS) will be summarized in a descriptive manner using Kaplan-Meier method including median and its 95% confidence interval (CI), progression rates and their 95% CI at 3 months, 6 month, 9 months, 12 months, and 15 months. In addition, Kaplan-Meier curves will also be presented for time-to-event variables.

The above efficacy data will be provided in listings.

## 7.5 Analysis of Safety Data

#### 7.5.1 Adverse Events

Adverse events will be classified into a standardized terminology MedDRA system organ classifications (SOC) and preferred terms (PT). Severity of AEs will be assessed by investigators according to CTCAE (v4.03).

A treatment-emergent AE (TEAE) will be defined as any new AE that begins, or any preexisting condition that worsens in severity during the treatment period, which is after the earlier date of first dose of niraparib, pembrolizumab or TSR-042 as applicable.

AEs that were possibly or definitely related to study drug niraparib or pembrolizumab or TSR-042 will be defined to be related to the study drugs while unrelated and unlikely related AEs will be defined as "not related". AEs with the closest relationship to study drugs will be used for summary.

Adverse events of special interest (AESI) will be collected and summarized.

- Patients who received pembrolizumab will be monitored for AESI caused by abnormal hepatic tests with an elevated AST or ALT value that is  $\geq 3 \times \text{ULN}$  concurrent with an elevated total bilirubin value that is  $\geq 2 \times \text{ULN}$  and, at the same time, an alkaline phosphatase value that is  $\leq 2 \times \text{ULN}$
- Patients who received niraparib will be monitored for
  - MDS and AML

- New malignancy information, i.e., any malignancy identified after the start of study medication
- o Pneumonitis
- o Embryo-fetal toxicity
- Regarding AESIs for TSR-042, no AESIs have been reported to date, therefore all serious AEs will be reasonably considered as AESI for patients who received TSR-042.

The number and percentage of patients who experienced an AE will be summarized. The denominator for calculating the percentages will be based on the number of patients in each cohort of the safety population.

The following types of summaries will be provided:

- Overview of TEAEs
- TEAEs by SOC and PT
- by SOC, PT, and Maximum CTCAE toxicity grade
  - o TEAE
  - o CTCAE Grade 3 or Greater TEAEs
- TEAEs by PT in descending frequency
- Drug-related TEAEs by SOC, PT, and Relationship to study drug
- by SOC, PT, Relationship to study drug, and Maximum CTCAE toxicity grade
  - o Drug-related TEAEs
  - o Drug-related CTCAE Grade 3 or Greater TEAEs
- by PT in descending frequency
  - o Drug-related TEAEs by PT in descending frequency
  - o Niraparib-related TEAEs by PT in descending frequency
  - o Pembrolizumab-related TEAEs by PT in descending frequency
  - o TSR-042-related TEAEs by PT in descending frequency
- Treatment emergent SAE by SOC and PT
- Drug-related treatment emergent SAE by SOC, PT, and Relationship to study drug
- TEAEs leading to study drug interruption, reduction, and discontinuation
  - TEAEs leading to study drug interruption by SOC, PT, and Interrupted Drug
  - o TEAEs leading to study drug reduction by SOC, PT, and Reduced Drug
  - TEAEs leading to study discontinuation by SOC, PT, and Discontinued Drug
- Drug-Related TEAEs leading to study drug discontinuation SOC, PT,

Relationship to Drug, and Discontinued Drug

- TEAEs leading to death by SOC and PT
- Most commonly reported TEAEs (i.e., those events reported by  $\geq 5\%$  of all patients

If a preferred term or system organ class was reported more than once for a patient, the patient would only be counted once in the incidence for that preferred term or system organ class.

In tabulation by severity (i.e., CTCAE toxicity grade),

- For a given preferred term, only the most severe preferred term for each patient will be included.
- For a given system organ class, only the most severe system organ class for each patient will be included.

All AEs will be provided in a data listing.

#### 7.5.2 Study Drug Exposure and Compliance

The following study drug exposure and compliance parameters will be summarized:

• Duration of study drug exposure in months is defined as

max(Date of last dose of niraparib + 1, Date of last dose of pembrolizumab + 21) — min(Date of first dose of niraparib, Date of first dose of pembrolizumab)

30.4375

- niraparib exposure parameters
  - o Duration of niraparib exposure in months defined as

- Number of cycles initiated as continuous variable
- o Number of cycles initiated as a categorical variable (1 cycle, 2 cycles, etc.)
- Number of patients with at least one dose escalation
- Number of patients with at least one dose interruption
- Number of patients with at least one dose reduction

- Number of patients with at least one missed dose
- Starting dose for niraparib
- Cumulative niraparib dosage (mg) received defined as sum of all niraparib dose received. This will be derived using pill count data (dispensed returned), whenever available. If the returned pill count data is not available for a particular cycle, the dosing data along with dosing modifications will be used to compute cumulative dose for that cycle.
- o Actual dose intensity (mg/day) for niraparib defined as

Cumulative niraparib dosage (mg) received # of cycle initated × # planned dosing days per cycle

o Intended dose intensity (mg/day) for niraparib defined as

Intended dose (mg) at first cycle × # of planned niraparib dosing days per cycle # planned dosing days per cycle

- pembrolizumab exposure parameters
  - o Duration of pembrolizumab exposure in months defined as

 $\frac{\text{Date of last dose of pembrolizumab} - \text{Date of first dose of pembrolizumab} + 21}{30.4375}$ 

- Cumulative pembrolizumab dosage (mg) received defined as sum of all pembrolizumab dose received
- o Actual dose intensity (mg/wk) for pembrolizumab defined as

Cumulative pembrolizumab dosage (mg) received

Duration of pembrolizumab exposure (wk)

o Intended dose intensity (mg/wk) for pembrolizumab defined as

$$\frac{200 \text{ (mg)}}{3 \text{ (wk)}} = 66.7 \text{ (mg/wk)}$$

o Relative dose intensity (%) for pembrolizumab defined as

 $\frac{\text{Actual dose intensity}}{\text{Intended dose intensity}} \times 100\%$ 

- TSR-042 exposure parameters
  - o Duration of TSR-042 exposure in months defined as

(Date of last dose of TSR042 — Date of first dose of TSR042 + 21) for the first cycles + (Date of last dose of TSR042 — Date of first dose of TSR042 + 42) for applicable Cycle 5 or later 30.4375

- Cumulative TSR-042 dosage (mg) received defined as sum of all TSR-042 dose received
- Actual dose intensity (mg/wk) for TSR-042 defined as

Cumulative TSR042 dosage (mg) received

Duration of TSR042 exposure (wk)

o Intended dose intensity (mg/wk) for TSR042 defined as

$$\frac{500 \text{ (mg)}}{3 \text{ (wk)}} (or \frac{1000 \text{ (mg)}}{6 \text{ (wk)}}) = 166.7 \text{ (mg/wk)}$$

o Relative dose intensity (%) for TSR-042 defined as

$$\frac{\text{Actual dose intensity}}{\text{Intended dose intensity}} \times 100\%$$

Study drug exposure parameters will be summarized using descriptive statistics. Details of study drug administration, dose modifications and duration of exposure will be listed.

#### 7.5.3 Clinical Laboratory Evaluations

Clinical laboratory assessments (CBC, serum chemistry, TSH, T3 or FT3, and FT4) will be summarized by visit in descriptive nature. Descriptive statistics will be provided for continuous laboratory data and associated change from baseline. Frequency distribution will be provided for categorical laboratory.

Baseline and post-baseline results will be converted to SI units and categorized as low, normal, or high relative to the normal range. Shift tables will be done by visit for each cohort.

In addition, the worst toxicity grades for selected laboratory tests as listed in Appendix B will be determined for each patient based on worst abnormal high and abnormal low lab values. The shift table from baseline CTCAE grade to the worst NCI CTC grade will be provided.

Corrected calcium will be derived using the following formula:

Corrected calcium (mmol/L) = 0.02\*(40 - normal albumin (g/L)) + serum calcium (mmol/L)

Unless otherwise specified, for frequency laboratory tables, the denominators for calculating the percentages will be based on the number of patients with non-missing values at each visit in the Safety population of each cohort.

For shift table from baseline to post-baseline visit, the denominators for calculating the percentages will be based on the number of patients with non-missing values at both baseline and each post-baseline analysis visit in the Safety population of each cohort.

Liver function tests post baseline will be summarized at any post baseline by the following categories.

- ALT  $\geq$  3×ULN, ALT  $\geq$  5×ULN, ALT  $\geq$  10×ULN, ALT  $\geq$  20×ULN
- AST  $\geq 3 \times ULN$ , AST  $\geq 5 \times ULN$ , AST  $\geq 10 \times ULN$ , AST  $\geq 20 \times ULN$
- (ALT or AST)  $\geq$  3×ULN, (ALT or AST)  $\geq$  5×ULN, (ALT or AST)  $\geq$  10×ULN, (ALT or AST)  $\geq$  20×ULN
- Total bilirubin  $\geq 2 \times ULN$
- Concurrent ALT  $\geq 3 \times ULN$  and total bilirubin  $\geq 2 \times ULN$
- Concurrent AST  $\geq 3 \times ULN$  and total bilirubin  $\geq 2 \times ULN$
- Concurrent (ALT or AST)  $\geq 3 \times ULN$  and total bilirubin  $\geq 2 \times ULN$
- Concurrent (ALT or AST)  $\geq$  3×ULN and total bilirubin  $\geq$  2×ULN and ALP > 2×ULN
- Potential Hy's law: Concurrent (ALT or AST)  $\geq$  3×ULN and total bilirubin  $\geq$  2×ULN and ALP  $\leq$  2×ULN or missing

Concurrent measurements are those occurring on the same date

Urinalysis is only collected at screening. The data will be provided in a listing. Other laboratory data will also be provided in data listings.

#### 7.5.4 Vital Signs

Vital signs (systolic and diastolic blood pressure, pulse, temperature, and weight) will be summarized by visit. Actual values and changes from baseline will be summarized at each visit. Baseline is defined as the last observation prior to start of the first dose of study drug(s).

#### 7.5.5 Electrocardiogram

ECG summaries will present frequency table analysis of ECG interpretation (normal vs abnormal - NCS, abnormal - CS) by stage and overall for baseline and end of treatment. The shift table from Baseline to end of treatment will also be provided.

A separate summary will be provided for ECG measurements including heart rate, PR interval, QT interval, RR interval, and QRS complex.

QTc will be used for the data analysis and interpretation. Commonly used techniques including Bazett's (QTcB) and Fridericia's (QTcF) methods are applied. QTcF will be used for the primary QT evaluation. A summary of the number and percentage of patients with QTc interval exceeding some predefined upper limit (e.g., >450 ms, >480 ms, >500 ms) will be provided. A summary of the number and percentage of patients with change from baseline in QTc interval exceeding some predefined upper limit (e.g., >30 ms, >60 ms) will be provided.

Furthermore, a summary will also provide the number and percentage of patients for

- 1. maximum post-baseline QRS interval  $\geq$  120 ms,
- 2. heart rate  $\leq$  50 bpm and decrease from baseline  $\geq$  20 bpm or  $\geq$  120 bpm and increase from baseline  $\geq$  20 bpm
- 3. PR interval >=220 ms and increase from baseline > 20 ms.

Detailed ECG results will be provided in a data listing.

#### 7.5.6 Physical Examinations

Physical examinations will be provided in a data listing only.

#### 7.5.7 ECOG Performance Status

Summary of ECOG performance status will present frequency distribution for each category. The denominators for calculating the percentages will be based on the number of patients without missing values.

Details on ECOG status will be provided in a data listing.

#### 8 DEFINITIONS AND CONVENTIONS FOR DATA HANDLING

As a general rule, missing data values are not imputed unless otherwise specified below and, in presentation of categorical variables, unknown and missing data may be presented as a separate category in some case and the denominator will include unknown or missing values as appropriate.

#### 8.1 Definition of Baseline

For all evaluations unless otherwise noted, baseline is defined as the most recent measurement prior to the first administration of study drug. Baseline can be the same date as first dose, given the measurement is expected prior to first dose when only date information is available.

## 8.2 Analysis Visit Window

For safety parameters including clinical laboratory data, measurements collected from unscheduled visits will not be included in the by-visit summary tables but will be included in the listings.

## 8.3 Efficacy Data Handling

See Section 4.1

## 8.4 Safety Data Handling

For all safety data, only observed data will be used for analyses, and missing data will not be imputed.

## 8.4.1 Handling of Repeated Clinical Laboratory Tests

The last repeat of laboratory results will be used in the summary tables for that visit. All the laboratory test results (original test results and repeated results) will be included in the data listings.

## 8.4.2 Handling of Partial Dates for AEs

When determining the treatment emergent AE, partial dates will be handled as follows.

- If the day of the month is missing, the onset day will be set to the first day of the month unless it is the same month and year as study treatment. In this case, the onset date will be assumed to be the date of treatment.
- If the onset day and month are both missing, the month and day will be assumed to be January 1 unless the event occurred in the same year as the study treatment. In this case, the event onset will be set to the day of treatment to conservatively report the event as treatment-emergent.
- A completely missing onset date will be set as the day of treatment. If the resulting onset date is after a reported date of resolution, the onset date will be set equal to the date of resolution.
- Imputation of partial dates is used only to determine whether an event is treatmentemergent; data listings will present the partial date as recorded in the eCRF.

## 8.4.3 Handling of Partial Dates for Medications

A medication with a completely missing start date will be considered a prior medication. A medication with a completely missing stop date will be considered a concomitant medication.

When determining prior or concomitant medications, partial start dates of prior and concomitant medications will be assumed to be the earliest possible date consistent with the partial date. Partial stop dates of prior and concomitant medications will be assumed to be the latest possible date consistent with the partial date. In the case of completely missing stop date, medication will be assumed to be ongoing. In the case of complete missing start date, medication will be assumed to be prior medication.

# 9 REFERENCE

Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989;10(1):1-10.

#### 10 APPENDICES

# Appendix A. Response Criteria by Response Evaluation Criteria in Solid Tumors (RECIST), v1.1

#### **Evaluation of Target Lesions**

**Complete Response (CR):** Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.

**Partial Response (PR):** At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

**Progressive Disease (PD):** At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions.)

**Stable Disease (SD):** Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

#### **Evaluation of Non-Target Lesions**

**Complete Response (CR):** Disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes must be nonpathological in size (< 10 mm short axis).

Note: If tumor markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response.

**Non-CR/Non-PD:** Persistence of 1 or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits.

**Progressive Disease (PD):** Appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.

Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or Investigator).

#### **Evaluation of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

Table 8: RECIST Response for Patients with Measurable Disease

| Target Lesions | Non-Target Lesions | New Lesions | Overall<br>Response | Best Overall Response<br>when Confirmation is<br>Required* |
|---|---|---|---|---|
| CR | CR | No | CR | > 4 weeks Confirmation** |
| CR | Non-CR/Non-PD | No | PR | > 4 weeks Confirmation** |
| CR | Not evaluated | No | PR | |
| PR | Non-CR/Non-PD/Not evaluated | No | PR | |
| SD | Non-CR/Non-PD/Not evaluated | No | SD | Documented at least once > 4 weeks from baseline** |
| PD | Any | Yes or No | PD | No prior SD, PR, or CR |
| Any | PD*** | Yes or No | PD | |
| Any | Any | Yes | PD | |

Abbreviations: CR = complete response; PD = progressive disease; PR = partial response; RECIST = Response Evaluation Criteria in Solid Tumors; SD = stable disease

Note: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment.

<sup>\*</sup> See RECIST v1.1 publication for further details on what is evidence of a new lesion.

<sup>\*\*</sup> Only for nonrandomized trials with response as primary endpoint.

<sup>\*\*\*</sup> In exceptional circumstances, unequivocal progression in nontarget lesions may be accepted as disease progression.

# Appendix B. Common Terminology Criteria for Adverse Events v4.03 (CTCAE)

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which |
|---|
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |

| are protected by third party copyright laws and therefore have been excluded. |
|---|